CLINICAL TRIAL: NCT00786461
Title: The Treatment of Bartholin´s Cyst or Abscess With Silver Nitrate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Pinar Bor, M.D, Randers Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-000494-22
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Bartholin´s Cyst
Keywords: silver nitrate; marsupialisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: silver nitrate application to the Bartholin´s cyst — 5 mm in diameter and 5 mm in length crystalloid silver nitrate stick is inserted into the cyst or abscess cavity.
Procedure: silver nitrat stick — The silver nitrate treatment is performed under local anaesthesia on an outpatient basis. A simple vertical incision 1 cm in length is made in the vaginal mucosa and the underlying cyst or abscess wall. A crystalloid silver nitrate stick of 5 mm in diameter and 5 mm in length is inserted into the cyst or abscess cavity.

SUMMARY:
Silver nitrate treatment of Bartholin's cyst or abscess will be compared to marsupialization treatment.

It is expected that silver nitrate treatment is effective, simple, inexpensive and the least anaesthetic requiring procedure, which can easily be carried out in the outpatient setting.

DETAILED DESCRIPTION:
Background and objective:

Bartholin gland cysts and abscesses are common problems in women of reproductive age. The traditional treatment of Bartholin´s cyst or abscess is marsupialization, which has disadvantages, such as pain of long duration, scarring, risk of general anaesthesia and risk of recurrence. In the present study we use silver nitrate in the treatment of Bartholin's cyst or abscess and compare to marsupialization. We expect lower healing time, lower recurrence rate and less pain with the silver nitrate treatment.

Methods and materials:

30 patients with Bartholin´s cyst or abscess will be investigated. It is prospective randomized study. The silver nitrate treatment is performed under local anaesthesia on an outpatient basis. A simple vertical incision 1 cm in length is made in the vaginal mucosa and the underlying cyst or abscess wall. A crystalloid silver nitrate stick of 5 mm in diameter and 5 mm in length is inserted into the cyst or abscess cavity.

The standard marsupialization treatment is performed under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Women with a age of 18-60 years
* Should read and understand Danish
* All women inclusive pregnant should have a Bartholins cyst or abscess

Exclusion Criteria:

* Subject who cannot give written informed consent

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Recidive of bartholin´s cyst or abscess and Dyspareunia after treatment | up to one year after treatment

SECONDARY OUTCOMES:
Wound healing, local burning, sequelae, hospitalisation time | 3-4 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Randers Central Hospital, Randers, Randers, Denmark